CLINICAL TRIAL: NCT01245179
Title: Phase I Study to Determine the Safety and Tolerability of Escalating Doses of Panobinostat (LBH589) in Patients With Sickle Cell Disease
Brief Title: Study of Panobinostat (LBH589) in Patients With Sickle Cell Disease
Acronym: LBH589
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abdullah Kutlar (Other)
Collaborators: Secura Bio, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Abdullah Kutlar, Professor of Medicine, Director of Augusta University Sickle Cell Center, Augusta University
Organization: Augusta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589BUS43T
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell anemia; sickle cell thalassemia; HDAC inhibitor; hemoglobin F; sickle beta thalassemia; Fetal Hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panobinostat (Experimental): All patients will receive Panobinostat at specified dose levels and dosing schedules.
  Interventions: Drug: panobinostat

INTERVENTIONS:
Drug: panobinostat — Panobinostat oral capsules taken THRICE WEEKLY (Monday, Wednesday, and Friday) for 12 weeks, exploring the following dosing regimens:
  1. 15 mg MWF 3 weeks on, 1 week off (if needed)
  2. 15 mg MWF every week (starting dose)
  3. 20 mg MWF 3 weeks on, 1 week off
  4. 20 mg MWF every week
  Other Names: LBH589; LBH589 lactate; FARYDAK®

SUMMARY:
The goal of this clinical research study is to find out about the safety and effects of a drug called panobinostat when given to adults with sickle cell disease. Panobinostat is a pan histone deacetylase (HDAC) inhibitor. HDAC inhibitors have been shown to significantly increase hemoglobin F induction, which is well documented to improve outcomes in sickle cell disease. HDAC inhibitors are also known to potently inhibit cell-specific inflammation, which is a primary contributor to the debilitating effects of sickle cell disease. Given the relevance of these mechanisms of action in SCD, panobinostat may prove to contribute significantly to the management of SCD patients, a population in critical need of further effective treatment options.

DETAILED DESCRIPTION:
This is a one-arm, open-label, Phase I, dose-escalation study of Panobinostat administered via different dosing schedules. In each schedule, this study is designed to determine the MTD (maximum tolerated dose) and DLT (dose limiting toxicities) of panobinostat as a single agent, and to characterize the safety and tolerability of panobinostat in adult patients with sickle cell disease who have failed to respond to hydroxyurea therapy (clinically or hematologically) or are intolerant of or refuse hydroxyurea therapy. The study consists of a Screening Phase, Treatment Phase, and Post-Treatment Follow-up.

Screening Phase:

Subjects will be screened for eligibility within 28 days of baseline visit (Day 1). Screening assessments will include informed consent, physical exam, vital signs (height, weight, blood pressure, heart rate, height, weight, and respirations), review of medical history, review of concomitant medications, 12-lead electrocardiogram (ECG), echocardiogram, and laboratory assessments. Screening laboratory assessments will include the following: CBC with differential, reticulocytes, complete chemistry panel, LDH, serum ferritin, thyroid function testing, Hb F percentage, F-cells, viral serology, urine albumin/creatinine ratio, and serum pregnancy in all females of childbearing potential. Approximately 15 ml (1 tablespoon) of blood will be collected at the screening visit.

Treatment Phase:

The Treatment Phase is twelve weeks in duration. Each subject will be assigned to a specified dose level and dosing schedule and will remain with the assigned regimen, if tolerated, throughout the twelve-week period. Patients at a given dosing regimen must complete at least 4 weeks of treatment before treatment decisions are made for subsequent participants. Regardless of specific dosing assignment, all subjects will take study drug thrice weekly (Monday, Wednesday, and Friday) throughout the duration of the 12-week treatment period.

The first three patients to enroll in the study will be assigned to a dose level of 15 mg panobinostat, with continuous thrice weekly treatment for the entire 12-week treatment period. Based on how well this regimen is tolerated, the next group of three subjects will either be assigned the same regimen or a reduced, intermittent schedule of three weeks on treatment followed by one week off.

Treatment decisions will continue accordingly, after each group of three subjects is treated with a given regimen. Six patients must be treated safely at a given dosing regimen before enrollment can advance to the next, higher level. Once the Maximum Tolerated Dose is determined, all subsequent patients will be enrolled to that regimen, with a total of up to 18 subjects enrolled. The four dosing regimens to be explored are:

1. 15 mg MWF 3 weeks on, 1 week off (only needed if starting regimen requires dose de-escalation)
2. 15 mg MWF every week (starting dose)
3. 20 mg MWF 3 weeks on, 1 week off
4. 20 mg MWF every week During the Treatment Phase, safety and efficacy assessments will be performed at specified times, and will include: physical examination, vital signs (weight, blood pressure, heart rate, height, weight, and respirations), adverse events assessment, ECG, quality of life questionnaire (ASCQMe), and laboratory assessments. Treatment Phase lab assessments are to be performed at specified visits and include CBC with differential, reticulocytes, complete chemistry panel, LDH, serum ferritin, Hb F percentage, F-cells, thyroid function testing, urine albumin/creatinine ratio, and urine pregnancy test for women of childbearing potential. Approximately 15 ml (3 teaspoons) of blood will be collected at each treatment visit. Every four weeks, an additional 5 ml of blood will be collected for inflammatory markers and protein biomarkers, for a total of 20 ml. On Day 1 (pre-treatment) and Day 85 (post-treatment), when additional samples are collected for genetic/ mechanistic studies, total volume collected is 25 ml.

Study drug will initially be dispensed at the baseline visit and every four weeks thereafter. Study drug accountability should be assessed at every visit. All baseline assessments will be completed prior to the first dose of study drug.

Follow-Up Phase:

A follow-up visit will be performed 4 weeks after end of treatment. Follow-up assessments will include: physical examination, vital signs, adverse events assessment, ECG, and laboratory assessments (CBC with differential, reticulocytes, complete chemistry panel, LDH, Hb F percentage, F-cells, and inflammatory markers). Approximately 15 ml (3 teaspoons) of blood will be collected at the follow-up visit.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients ages ≥ 18 years
2. Confirmed diagnosis of homozygous SS or S-β0Thalassemia
3. Intolerance to hydroxyurea therapy, refusal of hydroxyurea therapy, or failure to respond (refractoriness) to hydroxyurea therapy, either clinically or hematologically.
4. Clinically significant sickle cell disease as defined by:

   1. At least two hospitalizations over the past twelve months for any complication of sickle cell disease; or
   2. At least three pain crises over the past twelve months that last four or more hours and require a visit to a medical facility for treatment with oral or parenteral narcotics; or
   3. History of recurrent leg ulcers; or
   4. History of Acute Chest Syndrome within the past five years; or
   5. History of priapism requiring medical intervention within the past two years; or
   6. History of stroke (but not currently on a chronic blood transfusion regimen).
5. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
6. Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.

Exclusion Criteria

1. Use of agents that can induce Hb F within 60 days of Day 1 (i.e. hydroxyurea, butyrates, decitabine, 5-azacytidine, IMiDs®, or erythropoietin). Prior use of HDACi, including panobinostat, is not an exclusion criterion if discontinued > 60 days.
2. Patients who have had a vaso-occlusive crisis within the past 2 weeks that required treatment with parenteral medication.
3. Impairment of GI function or GI disease that may significantly alter the absorption of panobinostat (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
4. Patients on a chronic transfusion regimen, or any patient who has Hb A% > 20% from a recent transfusion
5. Any of the following laboratory abnormalities derived from the screening visit:

   * Absolute neutrophil count (ANC) < 1.5 x 109/L
   * Hemoglobin < 6 g/dl
   * Platelets < 100x 109/L
   * Serum creatinine >1.5 x Upper limits of normal (ULN)
   * AST and ALT > 2.5 x ULN
   * Serum total bilirubin > 10 mg/dL
   * Serum direct bilirubin > 1 mg/dL
   * Albumin <3.0 g/dl
   * Serum potassium < Lower limits of normal (LLN)
   * Total serum calcium [corrected for serum albumin] or ionized calcium <LLN
   * Serum magnesium < LLN
   * Serum phosphorus < LLN
6. Known impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * Left ventricular ejection fraction (LVEF) < lower limit of the institutional normal as determined by screening echocardiogram
   * Complete left bundle branch block
   * Obligate use of a cardiac pacemaker
   * Congenital long QT syndrome
   * History or presence of ventricular tachyarrhythmia
   * Presence of unstable atrial fibrillation (ventricular response > 100 bpm). Patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria.
   * Clinically significant resting bradycardia (< 50 bpm)
   * QTc > 470 msec on screening ECG
   * Right bundle branch block + left anterior hemiblock (bifasicular block)
   * Angina pectoris 3 months prior to starting study drug
   * Acute MI 3 months prior to starting study drug
   * Other clinically significant heart disease (e.g., CHF, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
7. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease) that could cause unacceptable safety risks or compromise compliance with the protocol
8. Patients who are currently receiving treatment with any study drug or have been on any study medications within the past 60 days.
9. Patients who have undergone major surgery 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
10. Women of child-bearing potential (WCBP) who are pregnant or breast feeding or who do not agree to use two methods of birth control, including a barrier method, if they are sexually active. WCBP, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test at screening and negative urine pregnancy test within 72 hours prior to starting study treatment. In addition, all sexually active WCBP must agree to use double method of contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method.
11. Male patients whose sexual partners are WCBP not using a double method of contraception during and 3 months after the end of treatment. Males must agree to use a condom during any sexual contact with WCBP during study drug treatment, during dose interruptions, and for 3 months after the end of treatment.
12. Known diagnosis of HIV infection, Hepatitis B; or acute/chronic, active Hepatitis C
13. Patients with a prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
14. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
15. Patients who are currently receiving treatment with certain prohibited medications and cannot either discontinue this treatment or switch to a different medication prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Days 1, 8, 15, 22, 29, 43, 57, 85, 113
  To determine the safety and dose limiting toxicities of escalating doses of oral panobinostat in sickle cell disease

SECONDARY OUTCOMES:
Secondary Outcome Measure | Days 1, 8, 15, 22, 29, 43, 53, 85, 113
  To determine the effect of escalating doses of oral panobinostat on the following parameters:
  I.Overall HbF percentage and F cells
  II. Change in total hemoglobin
  III. Effect on serum inflammation markers and cytokines (every 4 weeks)
  IV. Effect on quality of life as measured by ASCQMe questionnaire (pre- and post-treatment)
Define mechanisms of effect of panobinostat (Hb F induction and anti-inflammatory effects) and discover biomarkers of treatment response | Day 1 and Day 85
  I. Define epigenetic changes in the HBB locus mediated by panobinostat to reverse Hb F silencing in vivo
  II. Define the mechanism(s) of anti-inflammatory effects
  III. Determine the effect of panobinostat on RBC sickling
  IV. Perform an integrated bioinformatics analysis of histone acetylation and gene expression transcriptome of SCD patients treated with panobinostat

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Kutlar, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States